CLINICAL TRIAL: NCT06976112
Title: Effects of Lean Pork Intake on Endothelial Function and Vasomotor Symptoms in Perimenopausal Women
Brief Title: Impact of Lean Pork on Endothelial Function in Perimenopause
Acronym: LEAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: #PBRC 2024-066; NPB PR-006186 (Other: National Pork Board)
Record Dates: First submitted 2025-04-23; First posted 2025-05-16 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-05

CONDITIONS: Cardiovascular Outcome; Overweight and Obese Women; Perimenopausal Women; Vasomotor Symptoms (VMS)
Keywords: Perimenopause; Perimenopausal; Vasomotor Symptoms; VMS; Menopause; Cardiovascular Health; Blood pressure; Pork; Vegetarian
MeSH Terms: conditions — Overweight | interventions — Diet, Plant-Based

STUDY DESIGN:
Intervention Model Description: Single site randomized control trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcome assessments will be conducted by staff members who are masked to the participant's intervention group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pork Diet (Experimental): All participants will receive 7 days x 4 weeks of meals and snacks following a dietary pattern high in pork.
  Interventions: Behavioral: Pork Diet
- Plant Diet (Experimental): All participants will receive 7 days x 4 weeks of meals and snacks following a plant based diet.
  Interventions: Behavioral: Plant Diet

INTERVENTIONS:
Behavioral: Pork Diet — The diet will follow the Dietary Guidelines for Americans with 80% of the meat consumption per week being pork. Other animal protein (e.g., turkey, chicken, beef) will be minimized in the dietary plans (≤ 20%) so lean and processed pork are the primary protein source consumed. Within each day, ~80% of the daily pork intake will be fresh, unprocessed lean cuts (e.g., tenderloin, loin chops, sirloin roast, flank, and rump roast) and ~20% will be cured sources (e.g., Canadian bacon, pork sausage).
  Arms: Pork Diet
Behavioral: Plant Diet — The diet will be a Lacto-Ovo Vegetarian Diet following the Dietary Guidelines for Americans with no more than 21 oz per week of animal protein (e.g., eggs, cheese).
  Arms: Plant Diet

SUMMARY:
The goal of this study is to examine the impact of a diet high in fresh lean pork, compared to a plant-based diet, on cardiovascular function and vasomotor symptoms in perimenopausal women with overweight and obesity. The main questions it aims to answer are:

1. How does a diet high in pork, compared to a plant-based diet, affects blood lipids, endothelial function, and blood pressure?
2. How does a diet high in pork, compared to a plant-based diet, affects blood nitrate, cardiometabolic biomarkers, inflammatory biomarkers, and vasomotor symptoms?

Researchers will compare the diet high in pork to a plant-based diet to see if pork helps improve cardiovascular and mesopause symptoms.

Participants will:

* Consume both of the diets, each for 4 weeks, with a washout period between 2 and 6 weeks in between the diets trials
* Visit the clinic 5 times with weekly meal pick ups during the diet trials
* Undergo testing procedures including: weight and body composition, blood pressure and pulse, endothelial function using ultrasound of upper arm, microvascular blood flow, blood draws, physical activity measurements, and questionnaires.

DETAILED DESCRIPTION:
Investigators expect about 30 women will be enrolled in this study. The expected time in this study will be between 11 and 15 weeks.

Participants will consume both of the following diets, each for 4 weeks, with a washout period between 2 and 6 weeks in between the diets when participants will consume their usual diet. The diets will be consumed in random order. Participants will not be able to choose the order. Participants will receive 7 days of meals and snacks for 4 weeks for each diet.

* PORK Diet: A diet following the Dietary Guidelines for Americans with at least 80% of meat consumption being pork per week including tenderloin, loin chops, sirloin roast, flank, rump roast, and small amounts of Canadian bacon and pork sausage.
* PLANT Diet: A Lacto-Ovo Vegetarian diet following the Dietary Guidelines for Americans with no more than 21 oz. per week of animal protein including eggs and cheese.

ELIGIBILITY:
Inclusion Criteria:

* Are female
* Are between 40 and 55 years of age
* Have a BMI (a number calculated from participant height and weight) between 28 and45 kg/m2
* Are experiencing irregular menstrual cycles but have not gone longer than 12 consecutive months without a period
* Are experiencing severe vasomotor (menopause) symptoms
* Are doing less than 3 hours per week of structured exercise
* Have systolic blood pressure between 120 and 140 mmHg and/or diastolic blood pressure between 80 and 90 mmHg
* Have "sugary" hemoglobin called hemoglobin A1c less than or equal to 6.5%
* Are willing and able to refrain from using oral mouth wash for the duration of the study because the alcohol in mouth wash inhibits nitrate synthesis
* Are willing and able to comply with both the study diets
* Are willing to collect blood for future research
* Can read, speak, and understand English

Exclusion Criteria:

* Hysterectomy (partial or full) or oophorectomy
* Using hormone replacement therapy use and/or hormonal contraception use 6 months prior to study start
* Has systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥ 90 mmHg)
* Triglycerides ≥350 mg/dL, low-density lipoprotein cholesterol (LDL-C) ≥190 mg/dL, and/or taking a lipid-lowering medication -Diagnosed cardiovascular disease, diabetes (type 1 or 2), or endocrine- related disease (e.g. thyroid, PCOS), unstable gastrointestinal disease, kidney, liver, and/or pancreatic disease
* Diagnosed cancer (except skin cancer) in the last 5 years
* Taking >1 blood pressure medication and/or taking 1 blood pressure medication for <3 months
* Taking phosphodiesterase-5 inhibitors, anti-coagulants, corticosteroids, metformin, or insulin.
* Weight change ≥6.6 pounds in the past 3 months, actively trying to lose weight, or unwilling to remain weight stable throughout the study
* Current smoking or vaping, Binge and/or heavy drinker
* Food allergies or other reasons preventing consumption of study foods with both study diets

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — * Cisgender people identify with the gender that aligns with the sex they were assigned at birth.
  * Nonbinary people do not identify exclusively as a man or boy or as a woman or girl.
Enrollment: 30 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Change in Macrovascular Function | From the beginning of the diet period to the end of the diet period at 4 weeks.
  Macrovascular function will be measured by endothelial function. Investigators will use brachial artery flow mediated dilation (FMD) using ultrasound. Ultrasound images will be captured (Cardiovascular Suit 4, QUIPU, Pisa, Italy) at three time points 1) end-diastole for each cardiac cycle at baseline (~30 s), 2) during occlusion (~5 min), and 3) after occlusion (~5 min). The shear rate will be calculated for each cardiac cycle as 8 × mean blood velocity/ diameter, and the shear rate area under the curve from cuff release to peak diameter will be quantified as an index of the stimulus for FMD. The FMD values will be expressed as relative (%) changes from baseline to peak diameter and FMD/SRAUC will be corrected for shear rate (FMD/shear rate [SR] area under the curve [AUC]) in order to account for shear stress inter-individual variability.
Change in Microvascular Function | From the beginning of the diet period to the end of the diet period at 4 weeks.
  Microvascular blood flow will be assessed by near-infrared spectroscopy for oxygenated hemoglobin/myoglobin (O2Hb/O2Mb), deoxygenated hemoglobin/myoglobin (HHb/HMb), total hemoglobin/myoglobin (tHb/tMb), and tissue oxygen saturation (StO2, %)
Change in Blood Lipids | From the beginning of the diet period to the end of the diet period at 4 weeks.
  A blood lipid panel (total cholesterol, triglycerides, LDL, and HDL) will be performed at each outcome visit.

SECONDARY OUTCOMES:
Change in Total Score for Hot Flash Related Daily Interference Scale | From the beginning of the diet period to the end of the diet period at 4 weeks.
  The Hot Flash Related Daily Interference Scale (HFRDIS) is scored by summing responses to 10 items that assess how hot flashes interfere with daily activities such as work, social interactions, sleep, mood, and concentration. Each item is rated on a scale from 0 (do not interfere) to 10 (completely interfere), resulting in a total score ranging from 0 to 100. Higher scores indicate greater interference from hot flashes, with the scale providing a reliable measure of symptom impact on quality of life.
Change in Total Score for Menopause Rating Scale | From the beginning of the diet period to the end of the diet period at 4 weeks.
  The Menopause Rating Scale (MRS) consists of 11 items grouped into three subscales: somatic, psychological, and urogenital symptoms. Each symptom is rated from 0 (no symptoms) to 4 (very severe), with a total score ranging from 0 to 44. Subscale scores are calculated by summing the items within each domain, and higher scores reflect greater severity of menopausal symptoms.
Change in Total Score for Greene Climacteric Scale | From the beginning of the diet period to the end of the diet period at 4 weeks.
  The Greene Climacteric Scale includes 21 items measuring psychological, somatic, and vasomotor symptoms, plus one item assessing sexual interest. Each item is rated on a 4-point scale from 0 (not at all) to 3 (extremely), with higher total and subscale scores indicating greater symptom severity. Scores are calculated by summing item responses within each domain and across the entire scale.
Change in Blood Nitrates/Nitrites | From the beginning of the diet period to the end of the diet period at 4 weeks.
  Levels of nitrates/nitrites will be assessed from a blood draw.
Change in Insulin and Blood Glucose | From the beginning of the diet period to the end of the diet period at 4 weeks.
  Insulin and glucose will be evaluated from a fasting blood draw.
Change in Inflammation and Immune responses | From the beginning of the diet period to the end of the diet period at 4 weeks.
  ICAM, VCAM, VEGF, CRP, oxidized LDL, and interleukin-6 will be evaluated from a fasting blood draw.
Change in Blood Pressure | From the beginning of the diet period to the end of the diet period at 4 weeks.
  Blood Pressure will be measured using the Welch Allyn CEO297 manual sphygmomanometers.

CONTACTS AND LOCATIONS:
Overall Officials: Hannah E Cabre, PhD, RDN, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be protected under HIPAA